CLINICAL TRIAL: NCT04459273
Title: PET Biodistribution Study of 68Ga-FAPI-46 in Patients With Different Malignancies: An Exploratory Biodistribution Study With Histopathology Validation
Brief Title: Prospective Exploratory Study of FAPi PET/CT With Histopathology Validation in Patients With Various Cancers
Acronym: FAPI PET RDRC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-000630; NCI-2020-03766 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-08

CONDITIONS: Bladder Carcinoma; Cervical Carcinoma; Cholangiocarcinoma; Hematopoietic and Lymphoid Cell Neoplasm; Hepatocellular Carcinoma; Malignant Adrenal Gland Neoplasm; Malignant Brain Neoplasm; Malignant Pleural Neoplasm; Malignant Skin Neoplasm; Malignant Solid Neoplasm; Malignant Testicular Neoplasm; Malignant Thymus Neoplasm; Neuroendocrine Neoplasm; Thyroid Gland Carcinoma; Urothelial Carcinoma; Cancer of Unknown Primary Site
MeSH Terms: conditions — Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Cholangiocarcinoma; Hematologic Neoplasms; Carcinoma, Hepatocellular; Adrenal Gland Neoplasms; Brain Neoplasms; Skin Neoplasms; Testicular Neoplasms; Thymus Neoplasms; Neuroendocrine Tumors; Thyroid Neoplasms; Carcinoma, Transitional Cell; Neoplasms, Unknown Primary | interventions — FAPI-46; Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Basic science (68GA-FAPI-46 PET/CT) (Experimental): Patients receive 68Ga-FAPi-46 intravenously (IV), and then undergo PET/computed tomography (CT) over 20-90 minutes. On another day, patients receive 18F-FDG and then undergo PET/computed tomography (CT) according to standard of care procedures (if applicable).
  Interventions: Procedure: Computed Tomography; Drug: Gallium Ga 68 FAPi-46; Procedure: Positron Emission Tomography; Radiation: 18F-FDG

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Gallium Ga 68 FAPi-46 — Given IV
  Other Names: 68Ga-FAPi-46; Gallium-68-FAPi-46
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Radiation: 18F-FDG — Given IV
  Other Names: 18F-fluorodeoxyglucose

SUMMARY:
This exploratory study investigates how an imaging technique called 68Ga-FAPi-46 PET/CT can determine where and to which degree the FAPI tracer (68Ga-FAPi-46) accumulates in normal and cancer tissues in patients with cancer. Because some cancers take up 68Ga-FAPi-46 it can be seen with PET. FAP stands for Fibroblast Activation Protein. FAP is produced by cells that surround tumors (cancer associated fibroblasts). The function of FAP is not well understood but imaging studies have shown that FAP can be detected with FAPI PET/CT. Imaging FAP with FAPI PET/CT may in the future provide additional information about various cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To define the biodistribution of gallium Ga 68 fibroblast activation protein inhibitor (FAPi)-46 (68Ga-FAPi-46) in normal and cancer tissues of patients with various malignancies.

SECONDARY OBJECTIVES:

I. To evaluate the degree of 68Ga-FAPi-46 accumulation observed by positron emission tomography (PET) imaging as opposed to the amount of FAP in excised cancer tissue.

II. To assess the 68Ga-FAPI-46 biodistribution correlation with 18F-FDG biodistribution and to define the frequency of the following phenotypes (FAP+/ FDG+, FAP-/ FDG+, FAP+/ FDG-, FAP-/ FDG-)

EXPERIMENTAL OBJECTIVE:

To assess the correlation of 68Ga-FAPI-46 biodistribution with 68Ga-DOTATATE or 18F-DOPA (FDOPA), depending on the specific indication in patients who had them available

OUTLINE:

Patients receive 68Ga-FAPi-46 intravenously (IV), and then undergo PET/computed tomography (CT) over 20-90 minutes. On another day, patients receive 18F-FDG and then undergo PET/computed tomography (CT) according to standard of care procedures (if applicable).

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following cancer types:

  * Brain cancer
  * Bladder cancer
  * Urothelial cancer
  * Testicular cancer
  * Skin cancer
  * Thyroid cancer
  * Hepatocellular carcinoma
  * Cholangiocarcinoma
  * Thymus cancer
  * Pleural cancer
  * Cervical cancer
  * Adrenal cancer
  * Neuroendocrine tumors
  * Hematologic cancer
  * Cancer of Unkown Primary
* Patients who are scheduled to undergo surgical resection or tissue biopsy of the primary tumor and/or metastasis
* Patients are ≥ 18 years old at the time of the radiotracer administration.
* Patient can provide written informed consent
* Patient is able to remain still for duration of imaging procedure (up to one hour)

Exclusion Criteria:

* Patient is pregnant or nursing
* Patients with any new cancer therapy between the baseline PET/CT and the investigational FAPI PET/CT
* Patient has underlying disease which, based on the judgment of the investigator, might interfere with the collection of high quality data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Biodistribution of gallium 68Ga-FAPi-46 in normal and cancer tissues | At 20-90 minutes after injection]
  Will be quantified by mean and maximum standardized uptake values (SUVmean and SUVmax).

SECONDARY OUTCOMES:
68Ga-FAPi-46 accumulation observed by positron emission tomography (PET)/computed tomography (CT) | Up to year 2
  Will be correlated with FAP expression in surgically removed or biopsy derived tumor tissue.
68Ga-FAPI-46 biodistribution correlation with 18F-FDG biodistribution | up to 2 years
  2. To assess the 68Ga-FAPI-46 biodistribution correlation with 18F-FDG biodistribution and to define the frequency of the following phenotypes (FAP+/ FDG+, FAP-/ FDG+, FAP+/ FDG-, FAP-/ FDG-)

OTHER OUTCOMES:
To assess the 68Ga-FAPI-46 biodistribution correlation with other PET tracers | 60 minutes after tracer injection
  The other PET tracer biodistribution will be described by mean and maximum standardized uptake values (SUVmean and SUVmax). The SUV of FAPI PET and the other PET tracers will be tested for correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Calais, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States